CLINICAL TRIAL: NCT07001267
Title: Prospective Randomized Observer Blinded Single Center Study Comparing 90-day Functional Outcome in Patients Who Received Intravenous Propofol Infusion Versus Inhalational Sevoflurane for General Anesthesia During Mechanical Thrombectomy in Patients Who Suffered From Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Arun George, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161241
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke Patients
Keywords: Inhalation anesthesia; Intravenous anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- inhalational sevoflurane (Active Comparator): When treated for acute ischemic stroke, patient will receive inhalation sevoflurane as anesthesia
  Interventions: Procedure: Anesthesia drugs during the surgery
- intravenous propofol infusion (Active Comparator): When treated for acute ischemic stroke, patient will receive intravenous propofol infusion as anesthesia
  Interventions: Procedure: Anesthesia drugs during the surgery

INTERVENTIONS:
Procedure: Anesthesia drugs during the surgery — During treatment for acute ischemic stroke, patients will be given either inhalation or intravenous anesthesia.

SUMMARY:
This study is being done to compare outcomes after surgery for individuals who receive anesthesia through by inhaling medication and individuals who receive anesthesia intravenously by needle when experiencing treatment for their stroke. Currently very little is known about the outcomes for patients when comparing these two techniques of providing anesthesia during surgery. This study will provide information regarding outcomes that will help health care providers decide which technique will be better for patients

DETAILED DESCRIPTION:
According to the National Center for Health Statistics, stroke is a leading cause of disability and in 2021 the number five cause of death in the United States1. Endovascular thrombectomy for patients experiencing acute ischemic stroke from the occlusion of a larger cerebral vessel has become a mainstay of treatment.2 Patients undergoing thrombectomy have significantly reduced disability when compared to patients who do not receive this therapy. Several studies have compared outcomes of patients receiving local anesthesia only or sedation versus general anesthesia during endovascular thrombectomy treatment.3,4 While questions remain, current consensus is that when these procedures are done on patients under general anesthesia, there are higher rates of recanalization (opening of the occluded blood vessel) and improved functional recovery. Currently, less is known about the impact of the general anesthesia technique (inhalation vs. intravenous) on disability and functional outcomes in stroke patients.

Aim: The aim of this study is to compare functional outcomes and disability in patients undergoing endovascular thrombectomy for acute ischemic stroke under general anesthesia using a volatile inhalational versus total intravenous anesthesia (TIVA) technique. Hypothesis: We hypothesize that patients receiving total intravenous anesthesia will have better functional outcomes and less disability compared to those receiving volatile inhalational anesthesia as measured by the 90 day modified Rankin score and compared in both groups.

Background and Significance

ELIGIBILITY:
Inclusion Criteria:

* >18 years Acute ischemic stroke requiring endovascular treatment.

Exclusion Criteria:

* <18 years
* Pregnant patients
* Patients with malignant hyperthermia
* Allergies or any contraindications to either inhalational or intravenous agents
* Patients already on intravenous anesthetic infusions
* Prisoners
* Students and employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Independence at 90 days | From enrollment to 90 days after treatment
  The primary end point is functional independence at 90 days evaluated with the modified Rankin Scale (mRS). We plan to compare the functional recovery in 90 days in patients undergoing inhalational versus intravenous general anesthesia during mechanical thrombectomy using the modified Rankin score (mRS) in patients who suffered an acute ischemic stroke.
  (The mRS assesses a patient's functional independence or dependence after a stroke. Scores range from 0 (no symptoms) to 6 (death), with 0-2 indicating functional independence and 3-5 indicating dependence. A separate category of 6 is often added for patients who have died)

SECONDARY OUTCOMES:
Comparison of National Institutes of Health Stroke Scale (NIHSS) score | From enrollment to 90 days after treatment
  Comparison of National Institutes of Health Stroke Scale (NIHSS) score at presentation and at 90 days between study groups.
Thrombolysis in Cerebral Infarction (TICI) score | From enrollment to 90 days after treatment
  Thrombolysis in Cerebral Infarction (TICI) score comparison between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Arun George, MD, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: No